CLINICAL TRIAL: NCT03495427
Title: The Utility of PSMA-PET Imaging for Detecting Early Metastatic Prostate Cancer in Men With High GC Decipher® Test Scores: A Sub-aim of the VANDAAM Study (MCC #18523)
Brief Title: PSMA-PET Imaging for Detecting Early Metastatic Prostate Cancer in Men w/ High Decipher Test Scores
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-19291
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Recurrent Prostate Cancer
Keywords: radioactive diagnostic imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radioactive Diagnostic Imaging (Experimental): Participants will receive F-DCFPyL PSMA PET imaging annually for 4 years. An administered dose of 9 ± 1 mCi (333 ±37 MBq) F-DCFPyL Injection will be administered via an in-dwelling catheter placed in an antecubital vein or an equivalent venous access.
  Interventions: Drug: F-DCFPyL Injection; Diagnostic Test: PSMA PET

INTERVENTIONS:
Drug: F-DCFPyL Injection — F-DCFPyL Injection is a radioactive diagnostic imaging agent indicated for imaging of patients with recurrent prostate cancer.
  Other Names: Imaging agent
Diagnostic Test: PSMA PET — PSMA PET imaging (for men with high GC >0.45) will be done after 2 years post-treatment, then yearly up to 5 years.
  Other Names: Prostate-specific Membrane Antigen (PSMA); Positron Emission Tomography (PET)

SUMMARY:
This study will enroll 60 patients previously enrolled to MCC#18523, "A Validation Study on the Impact of Decipher® Testing on Treatment Recommendations in African-American and Non-African American Men with Prostate Cancer: (VANDAAM)" that had high risk Decipher test results (Decipher score >0.45). Patients with a high genomic classifier (GC) score at diagnosis will be approached for formal consenting for PSMA-PET imaging at 2 years post treatment.

DETAILED DESCRIPTION:
Normally, some patients with prostate cancer undergo imaging tests to determine the extent (spread) of their disease. These imaging tests often give good information, but not in all patients and not every time. This study deals with a new imaging test known as F-DCFPyL-Prostate-specific Membrane Antigen (PSMA) Positron Emission Tomography (PET), or F-DCFPyL-PSMA PET. The objective of this study is to evaluate safety and usefulness of using F-DCFPyL in detecting recurrent/metastatic prostate cancer. The F-DCFPyL PET imaging technique is used in some parts of the world but is not currently standard imaging care. Better understanding how this new imaging test performs in identifying recurrent/metastatic prostate cancer may lead to better management of prostate cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll 60 patients previously enrolled to MCC#18523, "A Validation Study on the Impact of Decipher® Testing on Treatment Recommendations in African-American and Non-African American Men with Prostate Cancer: (VANDAAM)" that had high risk Decipher test results (Decipher score >0.45).
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* Previously enrolled to MCC#18523
* Genomic Classifier (GC) testing successfully completed on biopsy and/or surgical specimen
* Decipher score from participation on the MCC#18523 study meets the criteria for high-risk (>0.45)
* Treated with radical prostatectomy (RP) or radiation therapy (RT) (+/- short-term androgen deprivation therapy (ADT)) with ≥2 years follow up
* Age > 18

Exclusion Criteria:

* No follow up information available post treatment
* Unable to undergo PET imaging due to pre-existing comorbidities and/or claustrophobia
* Administration of any radioisotope within 5 physical half-lives OR any IV X-ray contrast medium within 24 hours OR any high-density oral contrast medium (oral water contrast acceptable) within 5 days prior to study drug injection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Concordance (AUC) Between High Tumor GC Risk Score and Positive PSMA-PET Imaging Findings | Up to 5 years
  To estimate the concordance between tumor GC risk score and early metastatic disease using PSMA-PET imaging.

SECONDARY OUTCOMES:
Rate of Positive PSMA-PET Findings | Up to 5 years
  5-yr positive PSMA-PET findings in men with high GC score. At the end of the study (5 years), cumulative incidence of positive metastasis on PSMA-PET imaging will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kosj Yamoah, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States